CLINICAL TRIAL: NCT05337722
Title: A Smartphone Intervention for Pregnancy Smoking Cessation With Peer Support
Brief Title: App for Pregnancy Smoking Cessation With Peer Support
Acronym: SFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Babes-Bolyai University (Other); Wake Forest University Health Sciences (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Cristian Meghea, Associate Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21HD103039 (NIH)
Record Dates: First submitted 2021-08-26; First posted 2022-04-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Smoking Cessation; Tobacco Smoking
MeSH Terms: conditions — Smoking Cessation; Tobacco Smoking

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- App+fixed MI (Experimental): The participants will use the SFT2.0 app and receive a fixed number of 4 counseling video sessions during pregnancy up to 1-month postpartum.
  Interventions: Behavioral: SFT 2.0
- Adaptive app + as-needed MI (Experimental): The participants will use the SFT2.0 app and receive as-needed prenatal and postnatal video counseling sessions (between 1 and 10 sessions) during pregnancy up to 1-month postpartum.
  Interventions: Behavioral: SFT 2.0
- Control (Active Comparator): Participants will receive low dose prenatal and postnatal MI video counseling, defined as one prenatal session and one postnatal session.
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: SFT 2.0 — The SFT 2.0 intervention will include the use of the SFT 2.0 smoking cessation app, Motivational Interviewing (MI) counseling, and the support of a peer person
  Arms: Adaptive app + as-needed MI; App+fixed MI
Behavioral: Active control — Low dose prenatal and postnatal MI video counseling, defined as one prenatal session and one postnatal session
  Arms: Control

SUMMARY:
The objectives of this project are to develop, implement, and test the feasibility and effectiveness of an artificial intelligence adaptive mobile pregnancy tobacco cessation app-based intervention using deep tailoring and a self-nominated support person, and to build mHealth research capacity in Romania. The central hypothesis is that the intervention will show evidence of feasibility and effectiveness in increasing positive support, pregnancy cessation, and postnatal abstinence. The intervention is grounded in Self-Determination Theory (SDT) and Motivational Interviewing (MI), a counselling style that is effective in assisting people to quit smoking. The app will be novel in its use of the unique functionality of smartphones, use of reinforcement learning (RL) and deep tailoring to continuously adapt the intervention, the emphasis on increasing positive support, and the use of the app by both smoker and support person. The long-term goal of the research program is to use mHealth for smoking cessation leveraging the unique functionality of smartphones and to continue building mHealth research capacity and developing research networks in Central and Eastern Europe (CEE) and other LMICs.

Aim 1 (R21 phase). Develop and test the feasibility and acceptability of the SFT2.0 app-based mobile smoking cessation intervention with a support person during pregnancy and postpartum in Romania. Through a user-centered and iterative design the investigators will enhance the SFT1.0 app, deepen the tailoring, incorporate RL, expand the app for use by any support person, and test the intervention including the app and MI video counseling in a series of usability studies and a 12-week open trial (n=20).

Aim 2 (R33 phase). Test the SFT2.0 app-based smoking cessation intervention in a hybrid effectiveness and implementation randomized controlled trial. The investigators will randomize 375 pregnant smokers and their support persons to i) a fixed arm, including the SFT2.0 app for both, and fixed pre- and postnatal MI counseling; ii) an RL-adaptive arm, with the app continuously optimizing as-needed MI counseling; or iii) control group.

Aim 3 (R21 and R33 phases). Develop mHealth research capacity by enhancing individual and institutional research capabilities in Romania and expanding the existing international research network.

ELIGIBILITY:
Inclusion Criteria:

* age>=18
* pregnant
* user of regular cigarettes
* availability of Android phone with broadband data

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 790 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in smoking cessation | 3 and 6 months after birth
  7-day point biochemically verified prevalence of tobacco use
Change in postpartum abstinence | 3 and 6 months after birth
  Fewer than 5 cigarettes smoked since birth
Reach | 1 month after birth
  Proportion and representativeness (e.g., age, ethnicity) of dyads who enroll in each trial arm compared to each other and the general population of pregnant women in Romania
Adoption | 1 month after birth
  Proportion of participants who enroll in SFT2.0 by recruitment strategy
Implementation | 1 month after birth
  Participants frequency of overall SFT2.0 use and of the different app components
User engagement | 1 month after birth
  quality of the user experience when interacting with SFT2.0 measured using the four constructs of the User Engagement Scale short form: focused attention (e.g., The time I spent using SFT just slipped away), perceived usability (e.g., I was frustrated while using SFT), aesthetic appeal (e.g., SFT was attractive), and rewarding (e.g., Using SFT was worthwhile). Each construct includes 3 items (score 3-15) and can be treated as subscales or as a summary score of user engagement (4-60). An overall engagement score can be calculated by adding all of the items together and dividing by twelve. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: Undecided
While the investigators are undecided, potentially all non-identifying individual data may be shared with other researchers

REFERENCES:
- [Derived] Blaga OM, Dascal MD, Onisor A, Fratila T, Morar A, Mihu D, Iuhas CI, Caracostea G, Muresan D, Foley K, Resnicow K, Meghea CI. Smartphone intervention for pregnancy smoking cessation with peer support: the study protocol of the SmokeFree Together 2.0 (SFT 2.0) randomised controlled trial. BMJ Open. 2025 Mar 24;15(3):e100259. doi: 10.1136/bmjopen-2025-100259. PMID 40132847